CLINICAL TRIAL: NCT02789618
Title: A Pilot Study to Substantiate the Use of the Jay Sensitivity Sensor Probe by Correlating the Results With the Those of Yeaple Probe, Schiff Air Blast, Visual Analogue Scale (VAS) and Oral Health Impact Profile Questionnaire (OHIP)
Brief Title: A Pilot Study to Substantiate the Use of the Jay Sensitivity Sensor Probe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Pesquisa e Ensino em Saúde, Porto Allegre, Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ORL-SEN-2267
Record Dates: First submitted 2016-05-18; First posted 2016-06-03 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-05

CONDITIONS: Dentine Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Prorenin Receptor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A01 (Active Comparator): Toothpaste containing calcium silicate and Sodium Monofluorophosphate (1450ppm F) and a gel containing sodium fluoride (1450ppm F)
  Interventions: Other: A01
- B99 (Active Comparator): Toothpaste containing Stannous Fluoride and a dentinal bonding agent
  Interventions: Other: B99
- M89 (Placebo Comparator): Toothpaste containing sodium fluoride (1450ppm F)
  Interventions: Other: M89

INTERVENTIONS:
Other: A01 — Subjects will brush their teeth twice a day using their assigned toothpaste for 56 days. The gel will be applied in the evening of three consecutive days during the study time period
  Arms: A01
Other: B99 — Subjects will brush their teeth twice a day using their assigned toothpaste for 56 days. The bonding agent will be professional applied immediately prior to the clinical assessments.
  Arms: B99
Other: M89 — Subjects will brush their teeth twice a day using their assigned toothpaste for 56 days.
  Arms: M89

SUMMARY:
Subjects with at least two teeth with dentinal hypersensitivity and who meet the study criteria will be enrolled onto this double blind, randomised, parallel, controlled clinical trial. After enrolment, suitable subjects will use a fluoride toothpaste for 4 weeks (wash out period). Baseline dentine hypersensitivity assessments will be conducted using tactile stimuli, air blast, and VAS methods. Tactile methods of assessment will include use of the Yeaple Probe and the Jay Sensitivity Sensor probe. Air blast assessments will be conducted using the Schiff cold air sensitivity scale. The Oral Health Impact Profile (OHIP) questionnaire will be completed at four defined time points during the study. The baseline assessments will be conducted on the two teeth identified during the screening visit.

On completion of the baseline assessments, subjects will be randomly assigned to product. Dentinal hypersensitivity assessments will be repeated after 18, 28 and 56 days of product use.

ELIGIBILITY:
Inclusion Criteria:

* Willing and physically able to carry out all study procedures.
* Willing to give written informed consent and complete a medical history form.
* Have one hypersensitive tooth in two quadrants with exposed roots, which are anterior to the molars and demonstrate cervical erosion/abrasion or gingival recession, which have an air-blast hypersensitivity score of 2 or 3 on the Schiff sensitivity scale at Screening and a tactile hypersensitivity score of 10-60 grams of force using the Yeaple probe at baseline.
* Willing to comply with the oral hygiene and food and drink restrictions.

Exclusion Criteria:

Individuals with the following conditions will not be eligible for participation in the study:

* Subjects who have used anti sensitivity products in the 4 weeks prior to screening
* Subjects likely to require the use of professional dentinal desensitising therapy during the study.
* Subjects with an active oral ulcer (aphthous ulcer), or have similar experience within past 1 month.
* Subjects whose indicator teeth have abnormal oral pathology, for example:

  * Extensive restoration.
  * Observable caries.
  * Observable cracked enamel.
  * Leaking fillings or other restorations.
  * Cracked Tooth Syndrome
  * Suspected pulp pathology/abscess/pulpitis.
  * Atypical facial pain
  * Any tooth surface adjacent to those surfaces under investigation, which in the opinion of the investigator have any other condition(s) that provide confusing symptoms to those of cervical dentine hypersensitivity.
* Currently undergoing dental treatment, including orthodontic treatment.
* Subjects who had vital bleaching
* Investigational teeth are or are likely to become denture abutments during the course of the study.
* Known allergies to toothpaste and serum ingredients, including the flavour components.
* Obvious physical disability reducing tooth brushing ability.
* Receiving concomitant medication/therapy that might affect dentine hypersensitivity, e.g. regular use of analgesics, anti-histamines, SSRI medication
* Severe gingivitis, periodontitis and/or marked tooth mobility.
* Gingival surgery in the previous six months.
* Subjects with any serious concomitant diseases or medical or psychological conditions.
* In the opinion of the investigator unable to comply fully with the trial requirements.
* Participation in other dental clinical trials.
* Pregnant or breastfeeding (Self-Reported)
* Subjects who have participated in an oral care study within the previous 3 months.
* Diabetic (both Type 1 and Type 2)
* Previous history of rheumatic fever or heart valve pathology or require antibiotics for prophylaxis against bacterial endocarditis.
* Medical condition(s) and/or regular use of any medication, which either could affect the scientific validity of the study or if the subject was to participate in the study could, affect their wellbeing.
* Use of anticonvulsants; antihistamines; anti-depressants; sedatives; tranquilisers; anti-inflammatory drugs or daily analgesics.
* Full or removable partial dentures.
* The subject is an employee of Unilever or the site conducting the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Dentin hypersensitivity as measured using the Jay Probe | Baseline, 18 days, 29 days and 57 days
  Reduction in pain caused by dentin hypersensitivity will be measured using the Jay Probe (Tactile Stimulation) on day 18, day 29 and day 57 and compared to the baseline measurement
Dentin hypersensitivity as measured using the Yeaple Probe | Baseline, 18 days, 29 days and 57 days
  Reduction in pain caused by dentin hypersensitivity will be measured using the Yeaple Probe (Tactile Stimulation) on day 18, day 29 and day 57 and compared to the baseline measurement
Dentin hypersensitivity measured using the Schiff assessment | Baseline, 18 days, 29 days and 57 days
  Reduction in pain caused by dentin hypersensitivity will be measured using the Schiff assessment (Air Stimulation) on day 18, day 29 and day 57 and compared to the baseline measurement
An assessment of dentin hypersensitivity using the OHIP quality of life questionnaire | Baseline, 18 days, 29 days and 57 days
  Specific quality of life attributes and the impact of dentin hypersensitivity on subject's daily life will be measured (subjective measure)
Dentin hypersensitivity measured using the visual analogue scale (VAS) | Baseline, 18 days, 29 days and 57 days
  Reduction in pain caused by dentin hypersensitivity will be measured using the Visual Analogue Scale (VAS) on day 18, day 29 and day 57 and compared to the baseline measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Gomes, Principal Investigator — PENSA, Rua Carvalho Monteiro 234/601, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided